CLINICAL TRIAL: NCT03429725
Title: Increasing Individualism or Collectivism on Amazon Mechanical Turk Participants
Brief Title: Increasing Individualism and Collectivism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HSS-1502-P02-03
Record Dates: First submitted 2017-11-24; First posted 2018-02-12 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Individual Difference
MeSH Terms: interventions — Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualism (Experimental): Participant will be randomly allocated to either the individualism condition or the collectivism condition. For individualism condition, participant is tasked to write statements relating to his/her differences from the his/her immediate community, circle pronouns that relate to the self, and read passages related to individualism.
  Interventions: Other: Online prime (statements writing); Other: Online prime (circling); Other: Online prime (Sumarian Warrior); Other: Online prime (all)
- Collectivism (Experimental): Participant will be randomly allocated to either the individualism condition or the collectivism condition. For collectivism condition, participant is tasked to write statements relating to his/her similarities to the his/her immediate community, circle collective pronouns, and read passages related to collectivism.
  Interventions: Other: Online prime (statements writing); Other: Online prime (circling); Other: Online prime (Sumarian Warrior); Other: Online prime (all)

INTERVENTIONS:
Other: Online prime (statements writing) — Participants to write statements describing themselves or their similarities to their community.
Other: Online prime (circling) — Participants to circle either pronouns denoting themselves or pronouns denoting others.
Other: Online prime (Sumarian Warrior) — Participants read a passage which described the factors that led to his success in a war.
Other: Online prime (all) — Participants wrote statements, circled pronouns, as well as read the Sumarian Warrior passage.

SUMMARY:
An online survey is conducted on MTurk populations from India and USA. Participants were assigned either a condition with primes of individualism or one with primes of collectivism, before responding to a scale on culture and indicating details of their demographics.

ELIGIBILITY:
Inclusion Criteria:

* above age 21

Exclusion Criteria:

* below age 21
* not able to make decisions for self

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Higher collectivism or individualism level | 10 minutes
  Individualism and collectivism levels will be measured by Triandis & Gelfand (1998)'s "Culture Orientation Scale". This is a 16-item scale designed to measure: 1) Vertical Collectivism (VC) - seeing the self as a part of a collective and accepting hierarchy and inequality within that collective; 2) Vertical Individualism (VI) - seeing the self as fully autonomous, but recognizing and accepting the existence of inequality; 3) Horizontal Collectivism (HC) - seeing the self as part of a collective but viewing all the members of that collective as equal counterparts; and 4) Horizontal Individualism (HI) - seeing the self as fully autonomous, and believing in equality amongst individuals.
  All items are answered on a 5-point scale, ranging from 1= never or definitely no and 5 = always or definitely yes. Each dimension's items are summed up separately to create a VC, VI, HC, and HI score to reflect the level of collectivism and individualism in the sampled group.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale-NUS College, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided